CLINICAL TRIAL: NCT00666991
Title: A Phase 1 Study of Intraperitoneal Nanoparticle Paclitaxel in Patients With Peritoneal Malignancies
Brief Title: Pharmacokinetic, Safety and Efficacy Study of Nanoparticle Paclitaxel in Patients With Peritoneal Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CritiTech, Inc. (Industry)
Collaborators: University of Kansas Medical Center (Other); Beckloff Associates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC#11140; NCT00708864 (obsolete NCT alias)
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Peritoneal Neoplasms
Keywords: ovarian cancer; Mullerian tumors; peritoneal cavity carcinoma; gastrointestinal tract tumor; GI tract tumor; pancreatic cancer; colon cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Ovarian Neoplasms; Digestive System Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Nanotax, 50 mg/m2 (Experimental): Nanoparticulate paclitaxel (Nanotax) administered via intraperitoneal infusion at a dose of 50 mg/m2 once every 28 days until progression or unacceptable toxicity
  Interventions: Drug: nanoparticulate paclitaxel
- Nanotax, 82.5 mg/m2 (Experimental): Nanoparticulate paclitaxel (Nanotax) administered via intraperitoneal infusion at a dose of 82.5 mg/m2 once every 28 days until progression or unacceptable toxicity
  Interventions: Drug: nanoparticulate paclitaxel
- Nanotax, 125 mg/m2 (Experimental): Nanoparticulate paclitaxel (Nanotax) administered via intraperitoneal infusion at a dose of 125 mg/m2 once every 28 days until progression or unacceptable toxicity
  Interventions: Drug: nanoparticulate paclitaxel
- Nanotax, 175 mg/m2 (Experimental): Nanoparticulate paclitaxel (Nanotax) administered via intraperitoneal infusion at a dose of 175 mg/m2 once every 28 days until progression or unacceptable toxicity
  Interventions: Drug: nanoparticulate paclitaxel
- Nanotax, 225 mg/m2 (Experimental): Nanoparticulate paclitaxel (Nanotax) administered via intraperitoneal infusion at a dose of 225 mg/m2 once every 28 days until progression or unacceptable toxicity
  Interventions: Drug: nanoparticulate paclitaxel
- Nanotax 275 mg/m2 (Experimental): Nanoparticulate paclitaxel (Nanotax) administered via intraperitoneal infusion at a dose of 275 mg/m2 once every 28 days until progression or unacceptable toxicity
  Interventions: Drug: nanoparticulate paclitaxel

INTERVENTIONS:
Drug: nanoparticulate paclitaxel — This is a Phase 1, dose-escalation study with 6 cohorts of 1 - 6 patients. Patients receive Nanotax via intraperitoneal infusion once every 28 days continuing on this treatment schedule until disease progression or unacceptable toxicity is experienced. Dosing cohorts are as follows: 50 mg/m2, 82.5 mg/m2, 125 mg/m2, 175 mg/m2, 225 mg/m2, and 275 mg/m2.
  Other Names: Nanotax

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics and preliminary efficacy of an intraperitoneally administered suspension of nanoparticulate paclitaxel in patients with refractory malignancies principally confined to the peritoneal cavity.

DETAILED DESCRIPTION:
This is an open-label, Phase 1, dose-escalation study evaluating the safety, pharmacokinetics and preliminary efficacy of an intraperitoneally administered suspension of nanoparticle paclitaxel (Nanotax) in patients with refractory malignancies principally confined to the peritoneal cavity.

Nanotax will be administered via intraperitoneal infusion once every 28 days (equals one treatment cycle), continuing on this treatment schedule until disease progression or unacceptable toxicity is experienced.

This study will treat one patient per predefined dose level until one patient experiences a dose limiting toxicity (DLT) or until one patient has a Grade 2 or higher non-hematological toxicity or a Grade 3 or higher hematological toxicity during the first cycle of treatment. At this time, two additional patients will be treated at this dose level. If these 2 additional patients do not experience a DLT, then the next cohort of three patients will be treated at the next highest dose level. If 2/3 or 3/3 patients experience a DLT then the next cohort of three patients is enrolled at the next lower dose level. If 1/3 of the patients experience a DLT, then the next cohort of three patients is enrolled at the same dose level. If 0/3 patients experience a DLT, then the next cohort of three patients is enrolled at the next highest dose level. If 2 (or more)/6 patients at a given level experience a DLT, then the maximum tolerated dose has been exceeded and another cohort of three patients is treated at the next lower dose level.

The protocol will not treat above the highest dose level of 275 mg/m2.

Adverse event data will be collected throughout the study. Peritoneal fluid and blood samples will be collected prior to Nanotax administration and up to 14 days following infusion for Cycle 1 and Cycle 2 only. Evaluation of tumor response using RECIST criteria will be conducted following each treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age.
* Patients must have histologic or cytologic diagnosis of carcinoma predominantly confined to the peritoneal cavity.
* Patients must have failed all potentially curative therapy and have no other systemic treatment options available for extra-peritoneal disease. Patients with ovarian cancer that are platinum sensitive must have failed primary and at least one salvage regimen. Patients may undergo surgical debulking prior to entry into the trial.
* At least 28 days must have elapsed since completion of any other previous chemotherapy treatment received prior to registration in this study.
* Patients may have received prior abdominal surgery greater than 2 weeks prior to registration. Patients must have recovered from all effects of the surgical procedure.
* Patients must have a Zubrod Performance Status of 0 - 2.
* Patients must have a pretreatment granulocyte count greater than or equal to 1,500/microliter and platelet count greater than or equal to 100,000/microliter obtained within 14 days prior to registration.
* Patients must have adequate renal function as documented by a serum creatinine less than or equal to 1.5 times the institutional upper limit of normal obtained within 14 days prior to registration.
* Patients must have adequate hepatic function as documented by a bilirubin of less than or equal to 2 times the institutional upper limit of normal and an SGOT less than 5 times the institutional upper limit of normal obtained within 14 days prior to registration. Patients with hepatobiliary stents are eligible for this trial if the bilirubin meets the above parameter.
* There should be no plans for the patient to receive concomitant radiation therapy, hormonal therapy, or other chemotherapy for their tumor while on this protocol.

Exclusion Criteria:

* Patients with active inflammatory bowel disease or chronic diarrhea
* Patients with uncontrolled hypertension, unstable angina, symptomatic congestive heart failure, myocardial infarction within previous 6 months or serious uncontrolled cardiac arrhythmia
* Patients with active infection requiring systemic therapy
* Pregnant or nursing women
* Patients with Grade 2 or greater sensory neuropathy (by NCI Common Toxicity Criteria) at the time of study registration
* Patients taking concomitant medications demonstrated to inhibit or induce CYP3A4 or CYP2C8
* Patients with pre-existing conditions that prohibit the use of intravenous dexamethasone at the recommended dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose and to assess qualitative and quantitative toxicities | Through last patient visit

SECONDARY OUTCOMES:
Determine preliminary anti-tumor activity using RECIST criteria | Through last patient visit
Determine pharmacokinetics of intraperitoneal administration | Up to 14 days following Cycles 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Gary Johnson, M.D., Principal Investigator — University of Kansas Medical Center; Julia Chapman, M.D., Principal Investigator — University of Kansas Medical Center; Thomas K Schulz, M.D., Principal Investigator — Cancer Center of Kansas; Kathleen Moore, MD, Principal Investigator — Peggy and Charles Stephenson Oklahoma Cancer Center
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Peggy and Charles Stephenson Oklahoma Cancer Center, Oklahoma City, Oklahoma